CLINICAL TRIAL: NCT00757081
Title: Metabolic And Structural Effects Of Phosphatidylcholine And Deoxycholate Injections On Subcutaneous Fat
Brief Title: Study to Evaluate the Effect of Injection Lypolysis (Lipodissolve) Treatments to Reduce Body Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BodyAesthetic Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LD-001
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2009-05

CONDITIONS: Abdominal Subcutaneous Fat
MeSH Terms: interventions — Phosphatidylcholines; Deoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: phosphatidylcholine and deoxycholate

INTERVENTIONS:
Drug: phosphatidylcholine and deoxycholate — 50 mg phosphatidylcholine, 42 mg deoxycholate subcutaneous injection Every 8 weeks x 2 with additional 2 treatments optional
  Other Names: PPC; DC; Lipodissolve

SUMMARY:
The combination of phosphatidylcholine (PPC) and deoxycholate (DC) injected into subcutaneous fat is often popularly referred to as "Lipodissolve" therapy. Despite its attractiveness as an easy and noninvasive cosmetic treatment, the safety, effectiveness, and how the injections might work remain unclear. This study will investigate the hypothesis that injections of PPC/DC will reduce the amount body fat in the treated area. If so, the mechanisms responsible for the fat loss will be explored to find out whether fat cells die from toxic effects or are broken apart by the PPC/DC. Patients will receive at least 2 (no more than 4) treatments with PPC/DC injections every 2 months. Several methods of measuring fat loss will be used in the study, including photography and measurement of patients, tissue biopsy, blood tests, and MRI. The study will also record side effects of the treatments as well as patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* Body Mass Index (BMI) no greater than 30
* Excess fat in the lower abdomen area

Exclusion Criteria:

* Cigarette smoker
* Diabetes
* Pregnant or breast feeding
* Use anticoagulants (blood thinner), aspirin or other non-steroidal anti-inflammatory drugs that cannot be discontinued

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Subcutaneous fat thickness with calipers and MRI. | Before and 8 weeks after final treatment

CONTACTS AND LOCATIONS:
Overall Officials: V. Leroy Young, M.D., Principal Investigator — BodyAesthetic Research Center
Locations (1):
- BodyAesthetic Research Center, Creve Coeur, Missouri, United States

REFERENCES:
- [Derived] Reeds DN, Mohammed BS, Klein S, Boswell CB, Young VL. Metabolic and structural effects of phosphatidylcholine and deoxycholate injections on subcutaneous fat: a randomized, controlled trial. Aesthet Surg J. 2013 Mar;33(3):400-8. doi: 10.1177/1090820X13478630. Epub 2013 Feb 25. PMID 23439063
- See also: Related Info — http://www.bodyaesthetic.com